CLINICAL TRIAL: NCT02812875
Title: A Phase 1, Open-Label, Dose Escalation and Dose Expansion Trial Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Effects of Orally Administered CA-170 in Patients With Advanced Tumors and Lymphomas
Brief Title: A Study of CA-170 (Oral PD-L1, PD-L2 and VISTA Checkpoint Antagonist) in Patients With Advanced Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-170-101
Record Dates: First submitted 2016-06-14; First posted 2016-06-24 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Advanced Solid Tumors or Lymphomas
Keywords: Mesothelioma; PD-L1; VISTA; PD-1
MeSH Terms: conditions — Lymphoma; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CA-170 (Experimental): Taken orally in a once or twice daily schedule.
  Interventions: Drug: CA-170

INTERVENTIONS:
Drug: CA-170 — Dose escalation stage (Phase 1a) accelerated titration and standard 3+3 dose escalation in patients with advanced solid tumor or lymphoma.
  Dose expansion stage (Phase 1b) in patients with tumors that are shown to be responsive to anti-PD-1 or anti-PD-L1 checkpoint inhibitors and/or in tumor types known to express PD-L1 or VISTA, including but not limited to: mesothelioma, melanoma, non-small cell lung cancer, renal cell carcinoma, Hodgkin lymphoma, triple negative breast cancer, head and neck cancer, colorectal cancer, gastric cancer, bladder cancer, and ovarian cancer.

SUMMARY:
CA-170 is a rationally designed and orally available, small molecule that directly targets the Programmed death-ligands 1 and 2 (PD-L1/PD-L2), and V-domain Ig suppressor of T cell activation (VISTA) immune checkpoints and results in activation of T cell proliferation and cytokine production. This is a multi-center, open-label, Phase 1 trial of orally administered CA-170 in adult patients with advanced solid tumors or lymphomas who have progressed or are non-responsive to available therapies and for which no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age;
2. Life expectancy of at least 3 months;
3. ECOG PS ≤ 1;
4. Acceptable bone marrow and organ function at screening;
5. Ability to swallow and retain oral medications;
6. Negative serum pregnancy test in women of childbearing potential;
7. Measurable disease;
8. Tumor for which standard therapy, including approved anti-PD-1 or anti-PD-L1 therapy, when applicable, does not exist or is no longer effective. For patients enrolling into backfill of dose levels at or below the MTD/RP2D, patients with tumor types known to have a high VISTA expression (such as metastatic malignant pleural mesothelioma of epithelioid histology).

Exclusion Criteria:

1. Prior treatment anti-cancer therapy or use of any investigational agent within the past 28 days or 5 half-lives, whichever is shorter;
2. Toxicity from prior chemotherapy that has not resolved to Grade ≤ 1;
3. Radiotherapy within the last 21 days;
4. Primary brain tumors or CNS metastases;
5. Major or minor surgery < 28 and <14 days from the start of treatment, respectively;
6. Active autoimmune disease or any medical condition requiring the use of systemic immunosuppressive medications;
7. Endocrinopathies, unless on stable hormone replacement therapy;
8. Active infection requiring systemic therapy;
9. Receipt of live vaccines against infectious diseases within 28 days;
10. HIV positive or an AIDS-related illness;
11. Active/chronic HBV or HCV infection;
12. Uncontrolled CHF (NYHA Class 2-4), angina, MI, CVA, coronary/peripheral artery bypass graft surgery, TIA, or PE in prior 3 months;
13. Cardiac dysrhythmias;
14. Gastrointestinal disease that interferes with receipt of oral drugs;
15. Concomitant malignancy;
16. Pregnant or lactating female;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-05; Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
The number of patients with a dose-limiting toxicity (DLT) in the first treatment cycle | Approximately 24 months
Maximum tolerated dose (MTD) of CA-170 | Approximately 24 months
Recommended Phase 2 Dose (RP2D) of CA-170 | Approximately 24 months

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Profile of CA-170 | From Day 1 of Cycle 1(each cycle is 21 days)
  Maximum Concentration (Cmax)
Pharmacokinetic (PK) Profile of CA-170 | From Day 1 of Cycle 1(each cycle is 21 days)
  Area Under the Curve (AUC)
Preliminary Anti-tumor Activity of CA-170 based on RECIST and Immune Related Response Criterion (irRC) for Solid Tumors or Cheson for Lymphoma | 36 months

CONTACTS AND LOCATIONS:
Locations (20):
- United States (11):
  - University of California San Francisco, San Francisco, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Sarah Cannon Research Institute, Sarasota, Florida
  - Northwestern University, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Health System - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (3):
  - Hospital Clinic i Provincial, Barcelona
  - Catalan Institute of Oncology, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zong L, Mo S, Sun Z, Lu Z, Yu S, Chen J, Xiang Y. Analysis of the immune checkpoint V-domain Ig-containing suppressor of T-cell activation (VISTA) in endometrial cancer. Mod Pathol. 2022 Feb;35(2):266-273. doi: 10.1038/s41379-021-00901-y. Epub 2021 Sep 7. PMID 34493823
- [Derived] Li K, Tian H. Development of small-molecule immune checkpoint inhibitors of PD-1/PD-L1 as a new therapeutic strategy for tumour immunotherapy. J Drug Target. 2019 Mar;27(3):244-256. doi: 10.1080/1061186X.2018.1440400. Epub 2018 Feb 20. PMID 29448849